CLINICAL TRIAL: NCT02445742
Title: Single Nucleotide Polymorphism Association With Response and Toxic Effects in Patients With Ph+ CP-CML Treated With Bosutinib After Relapse to Previous Treatment
Brief Title: CML Treated With Bosutinib After Relapse
Acronym: BOSTRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOS-IIG-01
Record Dates: First submitted 2015-05-06; First posted 2015-05-15 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Chronic Myeloblastic Leukaemia
Keywords: Chronic Myeloblastic Leukaemia
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bosutinib (Experimental): 500 mg/day of Bosutinib during the study until disease progression, unacceptable toxicity, or withdrawal of consent occurs
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — 500 mg/day of Bosutinib during the study until disease progression, unacceptable toxicity, or withdrawal of consent occurs
  Other Names: Bostro

SUMMARY:
Prospective, open label, multicenter, phase II study evaluating correlation of SNPs with efficacy and toxicity in patients treated with Bosutinib. A total of 50 patients with previously treated Ph+ chronic phase CML will be included in the study

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form.
* Patients with chronic Ph + CML who presented a non-optimal response at 3 months prior to ITK treatment (imatinib, nilotinib, dasatinib). It is defined as a non-optimal response:

BCR-ABL> 10% per qRT-PCR (IS) at 3 months of initiation of treatment. BCR / ABL ≥ 1% per qRT-PCR (IS) at 6 months of initiation of treatment. BCR / ABL> 0.1% qRT-PCR (IS) at 12 months of initiation of treatment. BCR-ABL1> 0.1% qRT-PCR (IS) at any time after 12 months of treatment initiation.

* ECOG Performance Status of 0 or 1.
* Recovery at Grade 0-1, or at the baseline value of any pretreatment toxicity, except for alopecia. Cases with significant toxicity will be analyzed individually by the study coordinators
* Able to take daily oral capsules
* Adequate bone marrow function:

  1. Absolute neutrophil count > 1000/mm3 (>1000 x109/L)
  2. Platelets ≥ 100,000/mm3 (>100 x109/L)
  3. absent any platelet transfusions during the preceding 14 days.
* Adequate hepatic, and renal function:

  * AST/ALT ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 × ULN if attributable to liver involvement of leukemia
  * Total bilirubin ≤ 1.5 × ULN
  * Creatinine ≤ 1.5 × ULN
* Age > 18 years
* Willingness of male and female subjects, who are not surgically sterile or postmenopausal, to use reliable methods of birth control (oral contraceptives, intrauterine devices, or barrier methods used with a spermicide) for the duration of the study and for 30 days after the last dose of Bosutinib.

Exclusion Criteria

* Subjects with Philadelphia chromosome and bcr-abl negative CML.
* Overt leptomeningeal leukemia. Subjects must be free of CNS involvement for a minimum of 2 months. Subjects with symptoms of CNS involvement must have a diagnostic lumbar puncture prior to study enrollment.
* Subjects with extramedullary disease only.
* Prior stem cell transplantation.
* Major surgery within 14 days or radiotherapy within 7 days before the first dose of Bosutinib (recovery from any previous surgery should be complete before day 1)
* A history of a clinically significant ventricular arrhythmia, congenital or acquired prolonged QT interval, a baseline QTcF > 0.47 sec (average of triplicate readings) or unexplained syncope, uncontrolled or symptomatic congestive heart failure (CHF) within 3 months, or myocardial infarction (MI) within 6 months.
* Concomitant use of or need for medications known to prolong the QT interval
* Uncorrected hypomagnesemia or hypokalemia due to potential effects on the QT interval
* Recent (within 30 days of study entry) or ongoing clinically significant gastrointestinal disorder (e.g., malabsorption, short bowel syndrome, bleeding, or grade >1 diarrhea, nausea or emesis lasting more than 2 days, despite adequate medical therapy)
* Pregnant or breastfeeding women
* Evidence of serious active infection, or significant medical or psychiatric illness
* Known seropositivity to HIV, or current acute or chronic Hepatitis B or Hepatitis C (antigen positive), cirrhosis, hypokalemia (any grade), or clinically significant abnormal laboratory finding that would, in the investigator's judgment, make the subject inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Safety measured as adverse event gradation | 2 years
  Safety measured as graded adverse events described on common terminology criteria for adverse events

SECONDARY OUTCOMES:
Efficacy measured as response rate | 2 years
  Eficaccy measured as response rate to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luis Felipe Casado, Dr, Study Chair — PETHEMA Foundation
Locations (13):
- Spain (13):
  - C. H. U. de Gran Canaria Dr. Negrín, Gran Canaria
  - C. H. Gregorio Marañón, Madrid
  - C. U. La Paz - H. U. La Paz, Madrid
  - H. Ramón y Cajal, Madrid
  - H. U. de la Princesa, Madrid
  - H. U. Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - C. H. Regional de Málaga , H. General, Málaga
  - H. U. Son Espases, Palma de Mallorca
  - C. Asistencial U. de Salamanca, Salamanca
  - C. H. U. de Santiago, Santiago de Compostela
  - H. Virgen de la Salud, Toledo
  - Clínica Quirón Zaragoza S.A., Zaragoza